CLINICAL TRIAL: NCT06491654
Title: Effect of a Physiotherapy Program Based on Concurrent Strength and Moderate-to-high Intensity Aerobic Exercise Training, Along With Cohesive Bandaging, in Women With Breast Cancer-related Lymphedema.
Brief Title: Physiotherapy Program Impact on Breast Cancer-Related Lymphedema
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was discontinued because the estimated sample size necessary to obtain adequate statistical power was not reached.
Sponsor: European University Miguel de Cervantes (Other)
Collaborators: Hospital Clínico Universitario de Valladolid (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PI-DOC005-BCRL
Record Dates: First submitted 2024-02-22; First posted 2024-07-09 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Breast Cancer Related Lymphedema
Keywords: High-intensity functional training; Breast cancer; Lymphedema; Compression bandage; Strength exercise; Quality of life
MeSH Terms: conditions — Breast Cancer Lymphedema; Breast Neoplasms; Lymphedema

STUDY DESIGN:
Intervention Model Description: Prospective single-center randomized clinical trial.
Who Masked: Outcomes Assessor
Masking Description: The person analyzing the data collected (investigators, statisticians) will not know to which group each person belongs.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lymphedema experimental (Experimental): Subjects belonging to this group perform a 12-week supervised exercise. The patients will follow a moderate-to-high intensity strength exercise protocol, along with the application of a cohesive bandage (bandage will only be applied in subjects with Breast Cancer-Related Lymphedema, BCRL, and not in patients at risk).
  Interventions: Other: 12-week supervised exercise
- Healthy control (No Intervention): Subjects belonging to this group perform a 1-week supervised exercise, following the same training protocol as experimental group (arm 1). This group will not receive cohesive compressive bandage.

INTERVENTIONS:
Other: 12-week supervised exercise — During the study period (1 week for acute effects, 12 weeks for chronic effects), there will be 8 sessions per month, lasting 40-60 minutes each, with 2 sessions per week on alternate days, totaling 24 sessions. Each session includes: (1) warm-up (mobility exercises); (2) training: 5-min warm-up, followed by 15-min moderate-to-high intensity circuit of 7 functional global exercises with 10 reps each at a perceived exertion effort (RPE) of 5-7 on a scale of 1 to 10; (3) Aerobic exercise: starting at 15 mins, increasing by 5 mins biweekly to 30 mins by week 7; (4) Cool-down (general mobility); (5) Application of cohesive compressive bandage on the affected upper limb, worn for 2 hours post-session, removed at home. Participants may add a cotton bandage and finger bandage if needed.
  Arms: Lymphedema experimental

SUMMARY:
Breast Cancer Related Lymphedema (BCRL) is a sequela resulting from the application of certain treatments, such as axillary lymph node dissection and regional lymph node radiation. The main objective of the present clinical trial is to determine the effectiveness of moderate-high intensity strength training in combination with an aerobic exercise protocol and the application of cohesive compression bandaging in subjects with or at risk for BCRL and to analyze the acute responses of the molecular, functional and clinical profile of patients with BCRL or at risk after two sessions of intervention. To compare proteomic analysis of patients or at risk with healthy controls and to assess the adaptations produced after 12 weeks of exercise intervention and over a 12-week post-intervention period in patients with BCRL or at risk.

DETAILED DESCRIPTION:
Breast Cancer Related Lymphedema (BCRL) is a sequela resulting from the application of certain treatments, such as axillary lymph node dissection andregional lymph node radiation. Clinically, it can cause pain, swelling and a decrease in the functionality of those patients who suffer from it. Moderate-high intensity strength exercise, in combination with aerobic exercise and a cohesive compressive bandage, could minimize the associated symptomatology and clinical symptoms, as well as improve various biological parameters related to tumor progression and increase the functionality of patients. Likewise, the study of the long-term effects of the treatment will make it possible to determine the chronic adaptations generated by exercise.

The intervention will consist of concurrent training (strength and aerobic exercise) for all patients, whether they have BCRL or are at risk. Also, patients with BCRL will have cohesive bandaging applied at the end of the exercise session. The main objective of this study is to determine the benefits that moderate-high intensity strength training, in combination with an aerobic exercise protocol and, together with the application of a compressive bandage, generates on patients suffering from BCRL or at risk of suffering it. Through this investigation, we seek to analyze the impact of the intervention on various clinical, functional, and molecular factors. Likewise, healthy controls participants will participate in two exercise interventions and functional and molecular adaptations will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer survivors who have completed treatment (chemotherapy, surgery, and/or radiotherapy) at least 6 months prior to randomization for the trial.
* Patients diagnosed with unilateral stage I or II BCRL as established by the International Society of Lymphology Congress Working Group in 2020, or patients at risk of developing unilateral BCRL (who have received radiotherapy in the axillary region/radical mastectomy/modified radical mastectomy and lymph node dissection/breast surgery and sentinel lymph node biopsy).
* Age between 18 and 65 years.
* Voluntary participation in the study and informed consent.

Exclusion Criteria:

* Recent surgery (<3 months) or planned surgery during the study period.
* Patients with cognitive impairment.
* Patients with bilateral lymphedema.
* Health problems or illnesses that prevent them from participating in the intervention.
* Other serious conditions that may affect their HRQOL (Health-Related Quality of Life).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2024-03-11 (Actual); Primary Completion 2025-09-20 (Estimated); Study Completion 2025-10-10 (Estimated)

PRIMARY OUTCOMES:
Molecular variables: proteome. | 0 weeks, 1 weeks, 6 weeks, 12 weeks, 24 weeks.
  Venous blood samples are collected from the antecubital vein and kept at 4°C until preparation to avoid clotting and minimise protein degradation. Samples are centrifuged at 1500 g for 10 minutes at 4°C. Subsequently, the plasma is centrifuged at 2500g for 15 minutes at 4°C.
  Samples shall are stored at -80°C for subsequent analysis and only one freeze-thaw cycle shall be allowed. All samples shall are prepared within 1 hour of sample collection and show no signs of haemolysis.
  Likewise, a tear sample (5-15 µl) is taken from each eye, using a microcapillary for each eye. The sample is taken non-traumatically from the outer third of the tear meniscus. Samples are split and used both for cytokine analysis using a Luminex and frozen at -80°C for analysis.
  The protein concentration will be analyzed.
Functional variables: total session workload and total workload. | 0 weeks, 1 weeks, 6 weeks, 12 weeks, 24 weeks.
  The magnitude of the load is adjusted every 3 weeks to increase the intensity and volume of exercise.
  The number of repetition maxes and the peak force of these repetitions are recorded. Depending on the results obtained, the load is adjusted to 80% of the number of maximum repetitions or the intensity of the assigned rubber will be increased (when the number of repetitions is close to 20).
  The volume of aerobic exercise increases by 5 minutes every 2 weeks up to a maximum of 30 minutes.
Functional variables: physical activity levels | 0 weeks, 1 weeks, 6 weeks, 12 weeks, 24 weeks.
  Physical activity levels are recorded using an International Physical Activity Questionnaire (IPAQ). The results of the IPAQ indicate the METs/week of physical activity to classify the physical activity levels of each participant. The weighted MET-minutes per week (MET·min·wk-1) are calculated as duration × frequency per week × MET intensity, which are summed across activity domains to produce a weighted estimate of total physical activity from all reported activities per week (MET·min·wk-1).
  The items are structured to provide separate scores on walking; moderate-intensity; and vigorous-intensity activity as well as a combined total score to describe overall level of activity.
Functional variables: upper limb strength. | 0 weeks, 1 weeks, 6 weeks, 12 weeks, 24 weeks.
  To assess strength, a unilateral isometric test (chest press) is performed with a force sensor and 3 repetitions are performed with two minutes rest between repetitions for each upper limb. The peak force (N) of each isometric contraction is recorded.
Functional variables: lower limb strength. | 0 weeks, 1 weeks, 6 weeks, 12 weeks, 24 weeks.
  To assess strength, an isometric test (squat) is performed with a force sensor and 3 repetitions are performed with two minutes rest between repetitions. The peak force (N) of each isometric contraction is recorded.
Functional variables: manual grip strength. | 0 weeks, 1 weeks, 6 weeks, 12 weeks, 24 weeks.
  To assess strength, a manual grip strength test is performed with a hand-held dynamometer and 3 repetitions with three minutes rest between repetitions are performed for each upper limb. The peak force (kg) of each isometric contraction is recorded.
Functional variables: endurance and effort intensity | 0 weeks, 1 weeks, 6 weeks, 12 weeks, 24 weeks.
  Changes in measurements by a cycloergometer. Endurance and effort intensity is meadured in watts by a cycloergometer.
Functional variables: blood pressure | 0 weeks, 1 weeks, 6 weeks, 12 weeks, 24 weeks.
  Changes in systolic pressure and diastolic pressure in mm Hg.
Functional variables: gas consumption analysis | 0 weeks, 1 weeks, 6 weeks, 12 weeks, 24 weeks.
  Changes in oxygen consumption (VO2) and carbon dioxide production (CO2).
Functional variables: endurance and effort intensity. | 0 weeks, 1 weeks, 6 weeks, 12 weeks, 24 weeks.
  Changes in endurance and effort intensity in watts (W) measurements by a cycloergometer.
Functional variables: Heart rate. | 0 weeks, 1 weeks, 6 weeks, 12 weeks, 24 weeks.
  Changes in heart rate. Polar H10 Heart Rate Monitor with Chest Strap
Functional variables: Rate of perceived exertion (RPE) | 0 weeks, 1 weeks, 6 weeks, 12 weeks, 24 weeks.
  Changes in rate of perceived exertion (RPE). Using a numeric rating scale (NRS) of perceived exertion from 0 to 10 (known as the RPE CR-10 scale).
Functional variables: Electrical activity released by muscles by electromyography with surface electrodes to analyze muscle response. | 0 weeks, 1 weeks, 6 weeks, 12 weeks, 24 weeks.
  Changes in microvolts (µV).
Functional variables: Electrical activity released by muscles by electromyography with surface electrodes to analyze electrical activity. | 0 weeks, 1 weeks, 6 weeks, 12 weeks, 24 weeks.
  Changes in EMG frequency (Hz).
Health-related quality of life by Functional Assessment of Cancer Therapy Questionnaire for Breast Cancer (FACT-B and FACT-b+4). | 0 weeks, 6 weeks, 12 weeks, 24 weeks.
  The total FACT-G score consists of the sum of the four subdomains, ranging from 0 to 108. A higher score indicates a better Health-related quality of life (HRQoL).
Health-related quality of life by Upper Limb Lymphedema (ULL)-27 Questionnaire. | 0 weeks, 6 weeks, 12 weeks, 24 weeks.
  Upper Limb Lymphedema (ULL)-27:
  It is a scale that can describe all symptoms in one form, can provide a holistic approach, is easy to use, and can evaluate their ability to perform common functional activities in patients with Breast Cancer Related Lymphedema.
  The scale consists of 27 questions with physical, psychological, and social dimensions. 5-point Likert scoring scale (1 = strongly disagree, 5 = strongly agree) is used. The first 15 questions are on the physical dimension (min 15 and max 75 points), the questions between 16 and 22 on social dimension (min 7 and max 35 points), and the questions between 23 and 27 evaluate the social dimension (min 5 and max 25 points) of the individual. The total score of 27 questions is calculated for the global score. The lowest score is 27 and the highest score is 135 points. The high score of the scale shows that it affects the quality of life of the individual badly.
Disabilities of the Arm, Shoulder and Hand (DASH) Questionnaire. | 0 weeks, 6 weeks, 12 weeks, 24 weeks.
  Changes in total punctuation of questionnaire. The main part of the DASH is a 30-item disability/symptom scale concerning the patient's health status during the preceding week. The items ask about the degree of difficulty in performing different physical activities because of the arm, shoulder, or hand problem (21 items), the severity of each of the symptoms of pain, activity-related pain, tingling, weakness and stiffness (5 items), as well as the problem's impact on social activities, work, sleep, and self-image (4 items). Each item has five response options. The scores for all items are then used to calculate a scale score ranging from 0 (no disability) to 100 (most severe disability). The score for the disability/symptom scale is called the DASH score.
Numeric Rating Scale (NRS). | 0 weeks, 6 weeks, 12 weeks, 24 weeks.
  Numeric Rating Scale (NRS) typically consists of a series of numbers with verbal anchors representing the entire possible range of pain intensity. Generally, patients rate their pain from 0 to 10, from 0 to 20, or from 0 to 100. Zero represents "no pain," whereas 10, 20, or 100 represents the opposite end of the pain continuum (e.g., "the most intense pain imaginable," "pain as intense as it could be," "maximum pain").
Clinical variables: Blood pressure. | 0 weeks, 1 weeks, 12 weeks, 24 weeks.
  Changes in mean arterial pressure, systolic and diastolic pressure.
Clinical variables: Arm-ankle index | 0 weeks, 1 weeks, 12 weeks, 24 weeks.
  Changes in the measurements.
Clinical variables: Flow-mediated dilation of the brachial artery. | 0 weeks, 1 weeks, 12 weeks, 24 weeks.
  Changes in the measurements.
Clinical variables: Ankle-brachial index. | 0 weeks, 1 weeks, 12 weeks, 24 weeks.
  Changes in the measurements.
Clinical variables: Arm volume. | 0 weeks, 1 weeks, 12 weeks, 24 weeks.
  Changes in the measurements. Arm volume is calculated by making circumferences along the arm and converting them into volume (ml) using a truncated cone formula.
Clinical variables: Range of joint motion. | 0 weeks, 1 weeks, 12 weeks, 24 weeks.
  Changes in measurements (mean). The range of joint movement is calculated using a goniometer and the degrees of mobility are analysed.
Clinical variables: Heart rate variability. | 0 weeks, 1 weeks, 12 weeks, 24 weeks.
  Changes in heart rate monitoring. Heart rate variability is assessed by using a pulsometer and changes in variability are measured in the time interval between heartbeats.
Clinical variables: Ultrasound assessment of lymphedema. | 0 weeks, 1 weeks, 12 weeks, 24 weeks.
  Ultrasound assessment determines the thickness of subcutaneous and muscle tissue at different points of the upper limb: changes in thickness (in cm) will be assessed 10 cm distal and proximal to the elbow at the anterior, medial, posterior and lateral levels.
Clinical variables: Echocardiographic measurement. | 0 weeks, 1 weeks, 12 weeks, 24 weeks.
  Changes in functional cardiac modifications (left ventricular ejection fraction).
Clinical variables: Bone mineral density. | 0 weeks, 1 weeks, 12 weeks, 24 weeks.
  Changes in measurements by DXA (Dual-energy X-ray Absorptiometry).
Clinical variables: Body composition. | 0 weeks, 1 weeks, 12 weeks, 24 weeks.
  Changes in measurements by BMI (Body Mass Index) in kg/m^2.

CONTACTS AND LOCATIONS:
Overall Officials: Alejandro Santos Lozano, PhD, Principal Investigator — Universidad Europea Miguel de Cervantes
Locations (1):
- European University Miguel of Cervantes, Valladolid, Castille and León, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Executive Committee of the International Society of Lymphology. The diagnosis and treatment of peripheral lymphedema: 2020 Consensus Document of the International Society of Lymphology. Lymphology. 2020;53(1):3-19. PMID 32521126